CLINICAL TRIAL: NCT03174496
Title: Physical Activity Tracking in Paediatric Elective Tonsillectomy
Acronym: PATIPS
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Principal Investigator, Victoria Ziesenitz, MD, University Children's Hospital Basel
Other Study IDs: UKBB 2017-012; BASEC 2017-00547 (Other: Swissethics)
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Tonsillectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children aged 4-7 years
- Children and adolescents aged 8-16 years

SUMMARY:
This pilot study will investigate the feasibility of physical activity tracking in patients aged 4-16 years before and after elective tonsillectomy as an innovative tool in paediatric research. The participating patients will receive a wearable physical activity tracker (CE-certified) that will continuously measure the patients' physical activity before and after an elective tonsillectomy, in addition to their parents' documentation of their child's activity in a conventional diary.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 16 years old, in 2 subgroups (4-7 years, 8-16 years)
* Inpatient surgery at University Children's Hospital Basel (UKBB), Switzerland
* Children undergoing an elective tonsillectomy or tonsillotomy. Children having additional ENT procedures, such as adenectomy, tympanostomy, etc. may be included as well.

Exclusion Criteria:

* Children with mental or physical impairment during daily-life activities.
* Children undergoing additional surgical procedures other than Ear, Nose & Throat (ENT) procedures impacting the recovery period.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing elective tonsillectomy or tonsillotomy
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of physical activity tracking in children | up to 6 weeks
  Difference in proportions of patients having complete activity measurement data, comparing the electronic tracker with the conventional diary.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ziesenitz, MD, Principal Investigator — University Children's Hospital Basel
Locations (1):
- University Children's Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambrechtse P, Ziesenitz VC, Atkinson A, Bos EJ, Welzel T, Gilgen Y, Gurtler N, Heuscher S, Cohen AF, van den Anker JN. Monitoring the recovery time of children after tonsillectomy using commercial activity trackers. Eur J Pediatr. 2021 Feb;180(2):527-533. doi: 10.1007/s00431-020-03900-4. Epub 2021 Jan 4. PMID 33394138